CLINICAL TRIAL: NCT03989583
Title: Thermographic Analysis of Foot and Footwear in Children
Brief Title: Children´s Foot and Footwear Temperatures
Status: Completed | Type: Observational
Sponsor: Marina Fontán- Jiménez (Other)
Responsible Party: Sponsor-Investigator, Marina Fontán- Jiménez, Principal Investigator, Universidad de Extremadura
Organization: Universidad de Extremadura (Other)
Other Study IDs: UExtremadura
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Thermography
Keywords: Thermography; Children; Foot; Shoes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children's feet temperature: The thermal images were taken from 162 children who were 9- 10 years old in two schools in Mérida (Badajoz), Spain. Their parents or legal guardians were informed and signed an informed consent. All children were taken infrared images, so that skin temperature was evaluated, by dividing the thermograms in regions of interest in dorsal and plantar images of each foot. Shoes were divided into two regions of interest. The measures were taken in two different days: the first day, children wore school footwear and the second sports shoes.
  Interventions: Other: Infrared thermography

INTERVENTIONS:
Other: Infrared thermography — Temperature observation in foot and footwear in healthy children

SUMMARY:
This research aims to find thermal differences in foot in a group of children, detecting the most suitable footwear to acquire optimal foot temperature and taking into account that children in school age usually wear sports shoes instead of school shoes in most dimensions of daily life. It is assumed by general population that sports shoes increase sweating and provide less perspiration apart from biomechanical criteria, so for this reason the investigators are going to examine which thermal pattern offers each variety of footwear.

DETAILED DESCRIPTION:
Infrared thermal image allows detecting object´s temperature visually in a non-contact way. That makes the technique useful for different applications like in construction/ building, ecology, industry and medicine. Evolution of thermographic equipments makes it more accessible. It is a non- contact, non- invasive technique that helps researchers monitoring body temperature. So that, it is used to investigate ocular, liver, kidney and brain diseases, dental diagnosis, breast cancer detection or even sports injuries.

It is increasing the use of thermographic imaging in podiatry, so the main trials concerned to diabetes mellitus, vascular disorder or dermatological applications.

Nevertheless, there is little known about children´s foot temperature. Main studies are related to core temperature or variations in temperature among different parts of the body of enfants.

In consequence, the investigators found a lack of information related to such a significant topic, not only for podiatrists, but also for population in general.

ELIGIBILITY:
Inclusion Criteria:

* Healthy 9- 10 years old children

Exclusion Criteria:

* Vascular disease or another pathology that could interfere with thermal pattern of foot
* Wore sports shoes daily
* Used any kind of plantar orthoses, heels…
* Didn´t have correctly singed informed consent
* Wore sandals
* Had a bandaged feet

Ages: 9 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The thermal images were taken from 162 children who were 9- 10 years old in two schools in Mérida (Badajoz), Spain. Their parents or legal guardians were informed and signed an informed consent. All children were taken infrared images, so that skin temperature was evaluated, by dividing the thermograms in regions of interest in dorsal and plantar images of each foot. Shoes were divided into two regions of interest. The measures were taken in two different days: the first day, children wore school footwear and the second sports shoes.
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2017-05-23 (Actual); Study Completion 2017-05-23 (Actual)

PRIMARY OUTCOMES:
Infrared temperature | march, 30- may, 23 2017
  Foot and footwear temperature in children

CONTACTS AND LOCATIONS:
Overall Officials: Julián F García, Study Director — Universidad de Extremadura
Locations (1):
- Universidad de Extremadura, Plasencia, Cáceres, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fernández-Cuevas I, Marins JC, Gómez-Carmona P, García-Concepción MA, Arnaiz-Lastras J, Sillerro-Quintana M. Reliability and reproducibility of skin temperature of overweight subjects by an infrared thermography software designed for human beings. Thermology International. 2012; 22(3): 130-137
- [Background] Martínez E, Castillo A, Martínez I, Castellote M. Metodología para la intervención en elementos históricos: el caso de la espadaña del convento de Nuestra Señora de la Consolación (Alcalá de Henares-Madrid-España). Informes de la Construcción. 2013; 65(531): 359-366.
- [Background] Čoh M, Širok B. Use of the thermovision method in sport training. Physical Education and Sport. 2007; 5(1): 85-94.
- [Background] Lahiri BB, Bagavathiappan S, Jayakumar T, Philip J. Medical applications of infrared thermography: A review. Infrared Phys Technol. 2012 Jul;55(4):221-235. doi: 10.1016/j.infrared.2012.03.007. Epub 2012 Apr 13. PMID 32288544
- [Background] Ring E. The historical development of temperature measurement in medicine. Infrared Physics & Technology. 2007; 49(3): 297-301
- [Background] NG EYK. A review of thermography as promising non-invasive detection modality for breast tumor. International Journal of Thermal Sciences. 2009; 48(5): 849-859.
- [Background] Hildebrandt C, Raschner C, Ammer K. An overview of recent application of medical infrared thermography in sports medicine in Austria. Sensors (Basel). 2010;10(5):4700-15. doi: 10.3390/s100504700. Epub 2010 May 7. PMID 22399901
- [Background] Mori T, Nagase T, Takehara K, Oe M, Ohashi Y, Amemiya A, Noguchi H, Ueki K, Kadowaki T, Sanada H. Morphological pattern classification system for plantar thermography of patients with diabetes. J Diabetes Sci Technol. 2013 Sep 1;7(5):1102-12. doi: 10.1177/193229681300700502. PMID 24124935
- [Background] Nagase T, Sanada H, Takehara K, Oe M, Iizaka S, Ohashi Y, Oba M, Kadowaki T, Nakagami G. Variations of plantar thermographic patterns in normal controls and non-ulcer diabetic patients: novel classification using angiosome concept. J Plast Reconstr Aesthet Surg. 2011 Jul;64(7):860-6. doi: 10.1016/j.bjps.2010.12.003. Epub 2011 Jan 22. PMID 21257357
- [Background] Ring EFJ, Jung A, Zuber J, Rutowski P, Kalicki B, Bajwa U. Detecting fever in polish children by infrared thermography. En: 9th International conference of quantitative infrared thermography. Poland, 2008.
- [Background] Kolosovas-Machuca ES, Gonzalez FJ. Distribution of skin temperature in Mexican children. Skin Res Technol. 2011 Aug;17(3):326-31. doi: 10.1111/j.1600-0846.2011.00501.x. Epub 2011 Feb 22. PMID 21338404
- [Background] Ring EF, Ammer K. Infrared thermal imaging in medicine. Physiol Meas. 2012 Mar;33(3):R33-46. doi: 10.1088/0967-3334/33/3/R33. Epub 2012 Feb 28. PMID 22370242
- [Background] International Academy of Clinical Thermology (IACT) [Internet]. Redwood City, USA: IACT [citado 8 enero 2017]. Disponible desde: http://www.iact-org.org/professionals/thermog-guidelines.html